CLINICAL TRIAL: NCT02003053
Title: A Randomized, Controlled Trial of Inspiratory Muscle Training (IMT)in the ICU and CCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00022663
Record Dates: First submitted 2013-11-21; First posted 2013-12-06 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Critically Ill; Respiratory Failure
Keywords: Critically ill; intubated; safety; feasibility; inspiratory muscle training
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- IMT (Experimental): In the IMT group, inspiratory muscle training will start with 30% of MIP, for five minutes twice a day with increments of 10 % (absolute) everyday. Supplemental oxygen will be given as needed. The exercise will be done seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Interventions: Device: Inspiratory Muscle Trainer
- Sham (Sham Comparator): In the SHAM group, sham device will be used to train subjects 5 minutes twice a day, seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Interventions: Device: Inspiratory Muscle Trainer

INTERVENTIONS:
Device: Inspiratory Muscle Trainer

SUMMARY:
Inspiratory muscle training (IMT) is an intervention used with success in the outpatient setting within the COPD population. Use of IMT is also theoretically possible during mechanical ventilation. This study will will assess the feasibility and safety of the study of IMT in the patient population.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients.
* Must have passed spontaneuos brething trial screening but failed the trial itself.
* Potential subject must be able to perform atleast 5 minutes of spontaneous breathing trial.

Exclusion Criteria:

* Known neuromuscular disease
* Unstable cardiac ischemia
* Tracheostomized patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Morris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Inspiratory Muscle Training: In the IMT group, inspiratory muscle training will start with 30% of MIP, for five minutes twice a day with increments of 10 % (absolute) everyday. Supplemental oxygen will be given as needed. The exercise will be done seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Inspiratory Muscle Trainer
- Sham: In the SHAM group, sham device will be used to train subjects 5 minutes twice a day, seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Inspiratory Muscle Trainer
Period: Overall Study
Arm/Group | Inspiratory Muscle Training | Sham
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inpsiratory Muscle Training: In the IMT group, inspiratory muscle training will start with 30% of MIP, for five minutes twice a day with increments of 10 % (absolute) everyday. Supplemental oxygen will be given as needed. The exercise will be done seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Inspiratory Muscle Trainer
- Total: Total of all reporting groups
Arm/Group | Inpsiratory Muscle Training | Sham | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (16.9) | 54.33 (3.78) | 51.29 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — This data was not collected. | NA — This data was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — This data was not collected. | NA — This data was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility of Inspiratory Muscle Training
Description: The number of patients tolerating Inspiratory Muscle Training or Sham.
Time Frame: Baseline and until participant is extubated or discharged from the critical care unit (up to 1 month post-baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Inspiratory Muscle Training | Sham
Number analyzed (Participants) | 4 | 3
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient from the time of enrollment in the study until the patient was either extubated or discharged from the critical care unit, whichever occurred first (up to 1 month post-baseline).
Groups:
- Inspiratory Muscle Training Group: In the IMT group, inspiratory muscle training will start with 30% of MIP, for five minutes twice a day with increments of 10 % (absolute) everyday. Supplemental oxygen will be given as needed. The exercise will be done seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Inspiratory Muscle Trainer
- Sham Group: In the SHAM group, sham device will be used to train subjects 5 minutes twice a day, seven days a week until patient achieves liberation from mechanical ventilation or ICU/CCU discharge.
  Inspiratory Muscle Trainer
Arm/Group | Inspiratory Muscle Training Group | Sham Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes